CLINICAL TRIAL: NCT04505761
Title: The Usability, Feasibility, and Tolerability of Virtual Reality for Rehabilitation From COVID-19: An Explorative Study
Brief Title: The Usability, Feasibility, and Tolerability of Virtual Reality for Rehabilitation From COVID-19
Acronym: COVRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVRehab
Record Dates: First submitted 2020-07-03; First posted 2020-08-10 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus; Post Intensive Care Unit Syndrome
Keywords: Virtual Reality; Rehabilitation; Post-intensive care syndrome
MeSH Terms: conditions — Coronavirus Infections; postintensive care syndrome

STUDY DESIGN:
Intervention Model Description: Participants are asked to use Virtual Reality as an add-on to standard physiotherapy for revalidation after COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will receive Virtual Reality as an add-on to standard physiotherapy after COVID-19.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participants will use a Virtual Reality headset with a range of applications applicable for rehabilitation after COVID-19. Applications target physical, psychological, and cognitive rehabilitation. VR headset will be used for six weeks first at the physiotherapist's practice, and when possible, at home.

SUMMARY:
Patients who receive intensive care are known to be at high risk for physical, psychological, and cognitive impairments, a constellation known as PICS. COVID-19 patients are expected to have high chances of suffering from PICS (PICS-COV) as they frequently require several weeks of intensive care and traditional PICS preventive measures are virtually impossible due to infection control precautions, prone positioning, and deprivation of social contact. To prevent PICS after ICU discharge in COVID-19 patients, physical therapy is recommended. From recent but limited experience it appears that even patients with COVID-19 who have not been admitted to the ICU can suffer from impairments in the same domains and sometimes to a similar degree of severity. Also for these patient group rehabilitation seems warranted.

Yet, the resources needed to provide rehabilitation treatment to COVID-19 patients are inadequate because healthcare systems faced a shortage of high-quality treatment for these impairments already before the COVID-19 crisis emerged. Virtual Reality (VR) provides potential to healthcare practitioners to administer fast, temporary, and tailor-made rehabilitation services at a distance, and offers a solution to address the impending surge of demand for rehabilitation after COVID-19 infection. VR consists of a head mounted display (HMD) that can bring the user by computer-generated visuals into an immersive, realistic multi-sensory environment. Current VR technology is accessible, easy in use for a large audience, and safe in use. There already exist multiple VR applications for providing physical, psychological, and cognitive rehabilitation. These applications have been brought together in a VR suite for rehabilitation after COVID-19. Patients visiting a physiotherapist for rehabilitation from COVID-19 will be asked to participate in this study. They receive a VR HMD for training purposes. This study aims to understand the usability, feasibility, and tolerability of VR for rehabilitation after COVID-19, and to pilot the effectiveness of VR improving the physical ability, mental and cognitive status of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has had COVID-19.
2. Patient has an indication for physical therapy in the context of rehabilitation after COVID-19.
3. At the day of recruitment, the estimated length of the physical therapy is at least 3 weeks after inclusion.
4. Patient is willing and able to comply with the study protocol.
5. Patient is at least 16 years old on the day the informed consent form will be signed.
6. Patient can read and understand the Dutch language.

Exclusion Criteria:

1. The patient is participating in another study interfering with this study.
2. Patient has difficulties to handle virtual reality:

   1. Patient suffers from delirium or acute confusional state.
   2. Patient has (a history of) dementia, seizure, or epilepsy.
   3. Patient has severe hearing/visual impairment not corrected.
   4. The skin of the patient's head or face is not intact (for example head wounds, psoriasis, eczema).
3. Patient has a high risk of contamination with a therapy resistant micro-organism e.g. MRSA.
4. Patients suffers from severe anxiety or depression (HADS≥16).
5. Red flags (see Appendix 1).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview with 15 patients on their experiences of VR for rehabilitation from COVID-19. | Day 42
  At the end of the study, 15 patients will be interviewed about their experiences using VR for rehabilitation from COVID-19. The interview will be semi-structured, including questions on usability, tolerability and efficacy of VR according to the patients. The interviews will be recorded, written out and coded by means of grounded theory analysis in Atlas.ti. Themes and subthemes will be constructed.
Use of VR | Day 42
  By means of digital tracking in the VR goggles, we aim to understand what games are used most often by the participants.
Semi-structured interviews with physiotherapists on their experiences of VR for rehabilitation from COVID-19. | Day 42
  At the end of the study, 10 physiotherapists will be interviewed about their experiences using VR for rehabilitation from COVID-19. The interview will be semi-structured, including questions on usability, tolerability and efficacy of VR according to the physiotherapists. The interviews will be recorded, written out and coded by means of grounded theory analysis in Atlas.ti. Themes and subthemes will be constructed.

SECONDARY OUTCOMES:
Change in baseline performance test (guidelines KNGF) - Patient specific complaints. | Day 0, day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we use a baseline performance test as constructed by the COVID-19 recommendations (RL 2.0) as issued by the Royal Dutch Society for Physical Therapy (KNGF). Measurements will be done at the start of the intervention period and the end of the intervention period for tracking progress.
  The baseline performance test consists of several items of which the patient specific complaints is the first.
  Patient specific complaints refer to complaints the patients aim to improve by means of physiotherapy. Outcomes are qualitative outcomes.
Change in baseline performance test (guidelines KNGF) - 6 minute walk test | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we use a baseline performance test as constructed by the COVID-19 recommendations (RL 2.0) as issued by the Royal Dutch Society for Physical Therapy (KNGF). Measurements will be done at the start of the intervention period and the end of the intervention period for tracking progress.
  The baseline performance test consists of several items of which the 6 minute walk test is the second.
  The 6 minute walk test studies the physical capacity of a patient. We measure at day 0 how many meter a patient can walk in 6 minutes and compare this to the meters a patient is able to walk at day 42.
Change in baseline performance test (guidelines KNGF) - one-repetition maximum test | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we use a baseline performance test as constructed by the COVID-19 recommendations (RL 2.0) as issued by the Royal Dutch Society for Physical Therapy (KNGF). Measurements will be done at the start of the intervention period and the end of the intervention period for tracking progress.
  The baseline performance test consists of several items of which hand grip strength is the third.
  The hand grip strength is measured by the One-repetition maximum test which measures the amount of kg's a patient can grip at his peakforce. Measurements are done at day 0 and day 42 and compared.
Change in baseline performance test (guidelines KNGF) - 30 sec sit to stand | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we use a baseline performance test as constructed by the COVID-19 recommendations (RL 2.0) as issued by the Royal Dutch Society for Physical Therapy (KNGF). Measurements will be done at the start of the intervention period and the end of the intervention period for tracking progress.
  The baseline performance test consists of several items of which the 30 sec sit to stand test for lower extremities is the fourth.
  The 30 seconds sit to stand test is for testing leg strength and endurance. A patient has to do as many sit to stand exercises in 30 seconds. Measurements are done at day 0 and compared to day 42.
Change in baseline performance test (guidelines KNGF) - Borgscale for fatigue | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we use a baseline performance test as constructed by the COVID-19 recommendations (RL 2.0) as issued by the Royal Dutch Society for Physical Therapy (KNGF). Measurements will be done at the start of the intervention period and the end of the intervention period for tracking progress.
  The baseline performance test consists of several items of which the Borgscale for fatigue is the final item.
  The borgscale for fatigue is a numerical scale (1-10) to rate physical exertion and fatigue. Patients fill in the scale at day 0 and day 42. Results are compared.
Change in activities of daily life. | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves physical performance, we will as well measure change in activities of Daily Life. This questionnaire (ADL) measures the ease of participating in activities of daily life (ADL) of the patient. The questionnaire consists of 22 questions ranging from 0 (not at all) to 3 (easily autonomous). Maximum score is 63.
Change in HADS. | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves psychological rehabilitation, we will measure change in HADS. The HADS (Hospital Anxiety and Depression Scale) is used to measure change in psychological outcomes before and after the intervention period. Questionnaire consists out of 14 questions with answers ranging from 0 (often) to 3 (almost never). All questions are summed up to a total of 42 points.
Change in CFQ. | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves cognitive rehabilitation, we will use the CFQ. The CFQ (Cognitive Failure Questionnaire) is used to measure change in cognitive outcomes before and after the intervention period. Questionnaire consists out 25 questions ranging from 0 to 5. All questions are summed up to a total of 100 points.
Change in SF12. | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves quality of life, we will use the SF12. The SF12 questionnaire is used to measure change in quality of life before and after the intervention period.
  SF12: SF12 measures via different scaled questions eight concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. The first four items together form the physical health scale. The latter four items form the mental health scale. The higher the scores, the better the physical and mental health. Highest possible score: 56. Lowest possible score: 12.
Change in positive health. | Day 0, Day 42
  To investigate whether adding VR to rehabilitation (perceivably) improves quality of life, we will as well use the Positive Health questionnaire. The Positive Health questionnaire is used to measure change in quality of life before and after the intervention period.
  Positive Health:Positive health consists out of 42 statements separated in 6 categories: bodily functioning, mental functioning, spiritual dimension, quality of life, social participation, daily functioning. Each question should be rated with a 0 (worst) to a 10 (best). The higher the scores, the better the quality of life.

OTHER OUTCOMES:
Patient characteristics related to use of VR | Day 0
  Age, gender, education, employment, lifestyle, experience with technology - qualitative measures.

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, Principal Investigator — Radboud University Medical Center; Bart Staal, PT, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only upon asking.

REFERENCES:
- [Derived] Groenveld T, Achttien R, Smits M, de Vries M, van Heerde R, Staal B, van Goor H; COVID Rehab Group. Feasibility of Virtual Reality Exercises at Home for Post-COVID-19 Condition: Cohort Study. JMIR Rehabil Assist Technol. 2022 Aug 15;9(3):e36836. doi: 10.2196/36836. PMID 35858254